CLINICAL TRIAL: NCT04116346
Title: Comparison Between Fasting and no Fasting Before Interventional Coronary Intervention on the Occurrence of Adverse Events: Randomized Controlled Trial of Non-inferiority (TONIC)
Brief Title: Comparison Between Fasting and no Fasting Before Interventional Coronary Intervention on the Occurrence of Adverse Events
Acronym: TONIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: APHP190397
Record Dates: First submitted 2019-09-26; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Fasting; Cardiac Catheterization; Percutaneous Coronary Intervention
Keywords: Fasting; Cardiac Catheterization; Percutaneous coronary intervention
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Intervention Model Description: Our study is a prospective, monocentric, controlled, single-blind, randomized trial in two parallel arms
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigating physician performing the interventional procedure and evaluating the safety judgment criteria will not be informed of the patient's randomization arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting group (No Intervention): Fasting for both solids and fluids for up to 6 hours pre-procedure
- Non Fasting group (Experimental): Usual meal on the day of the procedure and allowed to drink as usual
  Interventions: Other: Oral intake allowed

INTERVENTIONS:
Other: Oral intake allowed — Oral intake (food and fluids) allowed up to the time of the procedure
  Arms: Non Fasting group

SUMMARY:
Traditionally, patients are asked to fast prior to invasive cardiac procedures. There exists neither clear evidence nor guidance about the benefits of this.

Hypothesis/Objective :

To show that allowing unrestricted oral intake before a coronary interventional procedure is not inferior to imposing a pre-procedural fasting period, in terms of adverse events, in patients requiring coronary angiography or a planned or semi-urgent percutaneous coronary intervention.

Method:

The study is a prospective, monocentric, controlled, single-blind, randomized trial in two parallel arms. The investigating physician performing the interventional procedure and evaluating the safety judgment criteria will not be informed of the patient's randomization arm. In order to keep the blind, the medical and paramedical staff of the interventional cardiology room will not inquire about the fasting status of patients included in the study.

Patients are randomized either to the pre-procedural fasting arm or to the absence of pre-procedural fasting.

* No intervention: Pre-procedural fasting is defined by the absence of ingestion of fluids or solid food for at least 6 hours before the examination.
* Experimental: free feeding and drinking until the procedure.

Patients are followed for 4 hours after the end of the procedure at the hospital for adverse events (vagal discomfort, nausea, vomiting or hypoglycaemia).

Then a follow-up will be done at day 7 after the procedure (by telephone for outpatients or discharged from the hospital and in the cardiology department for patients still hospitalized on D7) to look for the occurrence of acute renal failure or pneumonia

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years undergoing elective coronary angiography or angioplasty procedures
* Agreement to participate and signed informed consent after information
* Affiliation to Social Security System

Exclusion Criteria:

* Patient requiring fasting for another procedure
* Immediate coronary emergency (STEMI, very high risk NSTEMI)
* Patient under artificial nutrition
* Hemodynamic instability
* Patient under guardianship or curators
* Pregnant women, breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 736 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2022-12-07 (Estimated); Study Completion 2022-12-07 (Estimated)

PRIMARY OUTCOMES:
Adverse events linked to oral intake before cardiac procedure: vasovagal complications or nausea or vomiting or hypoglycemia | 4 hours
  * Vagal reaction is defined by the presence of at least two of the following criteria occurring during the procedure or closure of the arterial approach or during the post-procedural observation phase, in the absence of other explanations:
    * nausea / vomiting, skin paleness, sweating
    * decrease in systolic pressure <100mmHg (or 15% decrease in baseline if systolic blood pressure <100 mmHg baseline)
    * decrease in heart rate below 60 bpm (or more than 15% decrease if basal heart rate is below 60bpm) .
  * Nausea evaluated by interrogation; vomiting noted by the doctor or nurse
  * Hypoglycemia defined by the measurement of a glycemia lower than or equal to 0.70 mg / dL. This measurement is performed in the examination room at the beginning and end of the procedure on blood taken from the arterial sheath.

SECONDARY OUTCOMES:
Post procedural acute renal failure | 5 days
  Defined by a 25% increase in serum creatinine compared with basal level, or an increase in serum creatinine of more than 44 μmol/l in 3 days after injection of contrast medium
Post procedural aspiration pneumonia | 7 days
  - All patients will be contacted or reviewed in clinic to assess for chest infection

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, France

IPD SHARING:
Plan to Share IPD: No
data are own by Assistance Publique - Hôpitaux de Paris, please contact sponsor for further information